CLINICAL TRIAL: NCT02084407
Title: Induction of Pluripotent Stem Cells From Human Fibroblasts of DM1 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Myologie, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DM1-Fibroblasts
Record Dates: First submitted 2014-03-04; First posted 2014-03-12 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-03

CONDITIONS: DM1
Keywords: DM1; Cardiopathy; Adult
MeSH Terms: conditions — Heart Diseases | interventions — Restraint, Physical; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- DM1 subject with cardiopathy (Active Comparator): Clinical examination, Skin biopsy, Blood and urine sampling
  Interventions: Other: Clinical examination, skin biopsy, blood and urine sampling
- DM1 subject without cardiopathy (Active Comparator): Clinical examination, Skin biopsy, Blood and urine sampling
  Interventions: Other: Clinical examination, skin biopsy, blood and urine sampling
- Not DM1subject (Active Comparator): Clinical examination, Skin biopsy, Blood and urine sampling
  Interventions: Other: Clinical examination, skin biopsy, blood and urine sampling

INTERVENTIONS:
Other: Clinical examination, skin biopsy, blood and urine sampling

SUMMARY:
The objective of the study is the modelisation of human cardiomyocyts from pluripotent stem cells in order to study the cardiac alterations induced by CTG expansions.

ELIGIBILITY:
Inclusion Criteria for DM1 patient with cardiomyopathy:

* aged 20-50
* DM1 confirmed by molecular analysis
* Confirmed cardiomyopathy (infrahissiens conduction disorders)
* able to sign the consent form
* affiliated to european social security.

Inclusion Criteria for DM1 patient without cardiomyopathy

* aged 20-50
* DM1 confirmed by molecular analysis
* No cardiomyopathy (no infrahissiens conduction disorders or other trouble linked to DM1)
* able to sign the consent form
* affiliated to european social security.

Inclusion Criteria for controls

* aged over 18
* brother, sister, father or mother of the DM1 patient
* No DM1 confirmed by molecular analysis (CTG repetition under 38)
* No cardiac disorders.
* able to sign the consent form
* affiliated to european social security.

Exclusion Criteria:

* no pragnant or nursing women
* patient unable to understand informed consent
* patient under juridic protection

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Measure of DM1 alterations in human cardiomyocytes derived from induced pluripotent stem cells | At baseline

SECONDARY OUTCOMES:
Molecular changes in human DM1 cardiomyocytes expressing pathogenic CUGexp-RNA | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Servais, MD PhD, Principal Investigator — Institute of Myology
Locations (1):
- Institute of Myology, Paris, France